CLINICAL TRIAL: NCT03345043
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety and Immunogenicity of VAL-339851 in Healthy Subjects
Brief Title: Safety, Tolerability, and Immunogenicity of VAL-339851 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VAL-339851-P101
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Influenza
Keywords: VAL-339851; H7N9 antigen mRNA; Influenza vaccine; Moderna
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VAL-339851 (Experimental)
  Interventions: Biological: VAL-339851
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: VAL-339851 — Escalating dose levels
  Arms: VAL-339851
Other: Placebo — Saline
  Arms: Placebo

SUMMARY:
This clinical study will assess the safety, tolerability and immunogenicity of VAL-339851 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Agrees to comply with the study procedures and provides written informed consent
* 18 to 49 years of age
* Body mass index between 18 and 35 kg/m2
* Negative urine pregnancy test at the Screening visit and the day of each vaccination for females of childbearing potential.
* Female subjects must either be of non-childbearing potential or use acceptable methods of contraception from at least 3 weeks prior to enrollment and through the end of study visit
* In good health based on medical history, physical examination, vital sign measurements and laboratory safety tests performed prior to initial study vaccination
* Has access to a consistent and reliable means of telephone contact and agrees to stay in contact with the study site for the duration of the study

Exclusion Criteria:

* Any ongoing, symptomatic acute or chronic illness requiring medical or surgical care
* Administration of another investigational product within 60 days, or 5 half-lives, whichever is longer
* Participation in an investigational study involving lipid nanoparticles
* A history of hypersensitivity or serious reactions to previous influenza vaccinations
* History of Guillain-Barré Syndrome within 6 weeks following a previous influenza vaccine
* History of narcolepsy
* Administration of any licensed (inactivated or live) vaccines within 4 weeks before enrollment or plans to receive any vaccine within 12 weeks of the last study drug administration; receipt of any other avian H7N9 influenza vaccine at any time prior to or during the study is exclusionary
* Any known or suspected immunosuppressive condition, acquired or congenital, as determined by history and/or physical examination.
* Any chronic administration of immunosuppressant or other immune-modifying drugs within 6 months prior to administration of study vaccine
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
* Any acute disease at the time of enrollment
* Any significant disorder of coagulation requiring ongoing or intermittent treatment
* Active neoplastic disease or a history of any hematologic malignancy
* History of alcohol abuse or drug addiction within 1 year before the planned day of dose administration
* A positive test result for drugs of abuse or alcohol at screening or before the first dose administration
* Persons employed in a capacity that involves handling poultry or wild birds.
* The subject has any abnormality or permanent body art (eg, tattoo) that, in the opinion of the investigator, would obstruct the ability to observe local reactions at the injection site
* Any condition, that in the opinion of the Investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of the study results
* A positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies at screening
* Donation of blood or blood products > 450 mL within 30 days of dosing

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
Frequency of solicited AEs (local and systemic reactogenicity events) | 7 days following each dose administration
Frequency of unsolicited adverse events | 21 days following each dose administration
Frequency of serious adverse events (SAE), adverse events of special interest (AESI), medically-attended AEs, and new onset of chronic illness | One year after last dose administration

SECONDARY OUTCOMES:
Titers of hemagglutinin inhibition (HAI) and microneutralization antibodies in comparison with baseline sample | One year after last dose administration
Seroconversion rates in comparison to baseline samples | One year after last dose administration

CONTACTS AND LOCATIONS:
Locations (1):
- Miami Research Associates, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feldman RA, Fuhr R, Smolenov I, Mick Ribeiro A, Panther L, Watson M, Senn JJ, Smith M, Almarsson Ӧ, Pujar HS, Laska ME, Thompson J, Zaks T, Ciaramella G. mRNA vaccines against H10N8 and H7N9 influenza viruses of pandemic potential are immunogenic and well tolerated in healthy adults in phase 1 randomized clinical trials. Vaccine. 2019 May 31;37(25):3326-3334. doi: 10.1016/j.vaccine.2019.04.074. Epub 2019 May 10. PMID 31079849